CLINICAL TRIAL: NCT04467866
Title: A Randomized Controlled Trial of ride-on Car Training With a Standing Posture for Enhancing the Effectiveness of Locomotor Experience in Toddlers With Mild and Moderate Motor Delays
Brief Title: A Randomized Controlled Trial of ride-on Car Training and Locomotor Experience in Toddlers With Different Motor Delays
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOST 109-2314-B-182-032 -
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2022-03

CONDITIONS: Mobility Limitation
Keywords: toddlers with motor delays; modified ride-on cars; severity level; locomotor experience; mobility; psychosocial function
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ROC-Stand(Mild) group (Experimental): The participant's performance is indicative of the extent to which early power mobility training is feasible for 1 to 3 years old and diagnosed as mild motor delay. Parents/caregivers and occupational therapists will be responsible for ride-on car with standing posture training.
  Interventions: Behavioral: A Ride-on Car with a Standing Posture
- ROC-Stand(Mod) group (Experimental): The participant's performance is indicative of the extent to which early power mobility training is feasible for 1 to 3 years old and diagnosed as moderate motor delay. Parents/caregivers and occupational therapists will be responsible for ride-on car with standing posture training.
  Interventions: Behavioral: A Ride-on Car with a Standing Posture
- Control(Mild) group (Active Comparator): The participant's performance is indicative of the extent to which early power mobility training is feasible for 1 to 3 years old and diagnosed as mild motor delay. The other occupational therapist will be responsible for regular therapy.
  Interventions: Behavioral: Regular Therapy Program
- Control(Mod) group (Active Comparator): The participant's performance is indicative of the extent to which early power mobility training is feasible for 1 to 3 years old and diagnosed as moderate motor delay. The other occupational therapist will be responsible for regular therapy.
  Interventions: Behavioral: Regular Therapy Program

INTERVENTIONS:
Behavioral: A Ride-on Car with a Standing Posture — The 2-hour training session is composed of two 30-minute driving sessions and two 25-minute natural play sessions, with a 10-minute break. Every week's treatment program will be before planned and adjusted by the therapist and the caregivers through discussion and clinical observation of participant's performance in the previous session. Training will concentrate on building the concept of casual-effect on the switch and car motion, goal-oriented driving in a hospital, and upper limb use in functional tasks with driving and hand use in functional tasks for exploration in natural play session.
  Arms: ROC-Stand(Mild) group; ROC-Stand(Mod) group
Behavioral: Regular Therapy Program — The goals are to improve certain motor skills or psychosocial skills based on each participant's current developmental stage. The general propose of the training is to facilitate the developmental scales and improve mobility, socialization and upper limb use in functional tasks. Each participant will have the opportunity to walk on the hallway/public space and interact with the therapist and caregivers depending on his/her motor abilities.
  Arms: Control(Mild) group; Control(Mod) group

SUMMARY:
The three purposes of this study are: 1) to compare the effectiveness of the ROC-Stand training on mobility, psychosocial function and social looking with conventional therapy in toddlers with mild and moderate motor disabilities, 2) to compare the effectiveness of ROC-Stand training on body function level and environmental factors with conventional therapy in toddlers with mild and moderate motor disabilities, according to International Classification of Functioning, Disability and Health (ICF) levels, and 3) to determine the effects of ROC-Stand training on the relationship among social looking, caregiver-child interactions and mastery motivation in toddlers with mild and moderate motor disabilities.

Based on the power analysis from the preliminary results of the pilot study, the investigator will recruit 92 toddlers with motor delays and further assign them to either mild or moderate motor delays group. The participants in each group will be randomly assigned to either the ROC-Stand training program or conventional therapy(Control) program, resulting the following four training groups: the ROC-Stand(Mild) group (n=23), the ROC-Stand(Mod) group (n=23), Control(Mild) group (n=23), and Control(Mod) group (n=23). The whole study duration will be 24 weeks, including a 12-week intervention and a 12-week follow-up. All programs will include 120 minutes/per session, 2 sessions/per week. Participants will continue their regular therapy during the whole study. Standardized assessments are provided for a total three times, including the time before and after the intervention and in the end of the follow-up phase. The head-mounted cameras worn by the participants and caregivers will record the social looking and interaction behaviors for one 2-hour session/per week during intervention. Participants will also wear three accelerometers throughout the 2-hour training. Assessments include mobility, socialization, behavioral coding, body function, family perception and participation. The findings of this study will provide us some optimal, alternative ways to enhance locomotor experience depending on each child's and family's needs.

DETAILED DESCRIPTION:
Locomotor posture as upright can increase infants' visual availability of destinations and induce their motivation to interact and explore with environment. Using a modified ride-on car (ROC) with a standing posture (ROC-Stand) may result in the similar effects. Our previous world's first randomized controlled trial (RCT) manipulated the parameters of the ROC experience by increasing the demands of postural control during the course of locomotion. The initial findings were positive and inspiring. After an intensive 12-week training program, toddlers with motor delays in the ROC-Stand group had significant improvements in mobility and social function. Moreover, the ROC-Stand group tended to have the most improvements than the ROC-Sit and conventional therapy groups, including mobility, social function and mastery motivation. The ROC-Stand group also had the highest goal achievement scores. In addition, the pilot results of caregivers' perceptions showed over 80% of the caregivers involved in the ROC training programs had decreased concerns on children's motor and social development. Their expectations changed due to the observed improvements in children's movements, cognition, and motivation. The intensive 3-month ROC training program, particularly the standing one, was feasible and beneficial for toddlers with motor delays and their caregivers.

However, the severity level of motor delay should be considered in the early PMDs and require further investigation on the related treatment effects. Thus, a further study of toddlers with different severity levels of motor delays will provide us a full investigation on the effectiveness of ROC-Stand training on mobility, psychosocial function and locomotor experience. Moreover, the integration of information regarding the social looking behaviors, motor cost, caregiver-child interactions and caregivers' perceptions will be beneficial for clarifying the influences of these factors on the outcomes. The purpose of this study is to examine the effectiveness of ROC-Stand training on mobility, psychosocial function and social looking in toddlers with mild and moderate motor disabilities. To obtain the information of social looking and interactions with their caregivers, the investigator will use the lightweight, head-mounted action camera to record children's behaviors. Up to now, there is no ROC-related study applying this methodology to investigate the ecological validity in toddlers with motor delays. This design may help us to capture the novelty and variability of real-world locomotor experience regarding social looking, exploration and interactions.

The specific aims of this study are: 1) to compare the effectiveness of the ROC-Stand training on mobility, psychosocial function and social looking with conventional therapy in toddlers with mild and moderate motor delays, 2) to compare the effectiveness of ROC-Stand training on body function level and environmental factors with conventional therapy in toddlers with mild and moderate motor delays, according to the ICF, and 3) to determine the effects of ROC-Stand training on the relationship among social looking, caregiver-child interactions and mastery motivation in toddlers with mild and moderate motor delays.

Study Design: A randomized, multiple group pretest-posttest control group design will be applied. Four groups will be involved in this project: ride-on car training with a standing posture for toddlers with mild motor delays (ROC-Stand(Mild)), ride-on car training with a standing posture for toddlers with moderate motor delays (ROC-Stand(Mod)), conventional therapy for toddlers with mild motor delays (Control(Mild)) and conventional therapy for toddlers with moderate motor delays (Control(Mod)). The investigator will use stratified randomization. They will be arranged to one of the two groups based on the motor composite (MC) scores assessed by Bayley-III. Subsequently, the participants in each group will be randomly assigned to either the ROC-Stand training program or conventional therapy program by using a computer program (Research Randomizer Form www.randomizer.org). The study duration for each participant is 24 weeks, including a 12-week training phase (intervention) and a 12-week follow-up phase.

There will be 4 groups, including the ROC-Stand(Mild) group (23 toddlers), the ROC-Stand(Mod) group (23 toddlers), the Control(Mild) group (23 toddlers) and Control(Mod) group (23 toddlers). The age group of infants/preschool children is selected based on the previous studies of ROC training in young children with motor disabilities.

Recruitment: The children will be recruited from self-referrals, health care practitioners, or the hospitals in Taipei and Taoyuan, Taiwan where children with motor delays are receiving outpatient rehabilitation. Parents/guardians will obtain information about the study through the flyers and their therapists. When the research team contacts the parents, study will be explained and parents will receive a letter detailing the procedure and given an opportunity to ask questions. Parents/guardians will sign this informed consent form at the time of the first visit.

Procedure: Before randomization, the participants will receive pre-intervention measurements, including developmental assessments, the evaluations of environmental factors and self-developed questionnaires. The self-developed questionnaires were designed to examine parental perceptions on the training program and children's capabilities in the previous studies. The pretest and posttest developmental assessments and questionnaires will be completed in a testing room at Chang Gung University by a licensed occupational therapist who is blinded to the study purpose and not involved in the training programs. These assessments will occur on three occasions: before and after the 12-week training phase, i.e., intervention (T1 & T2) and the end of the 12-week follow-up phase (T3). After the pretest, participants will be randomly assigned into 4 groups and started the training programs in the university.

During the 12-week intervention, the locomotor experience of social looking behaviors and interactions for the four training groups will be videotaped by the head-mounted action cameras worn by the participants and the caregivers for one 2-hour session/per week at the university. In addition, participants will wear three accelerometers on their wrists and right hip to monitor the energy expenditure and activity counts during the intervention phase. An activity log used in the previous studies will also be applied in the 4 groups to record the training conditions and the caregiver's feedback on the training program every week during the 12-week intervention. The activity log will be mostly qualitative data that involves caregivers' descriptions. For the 12-week follow-up phase, all participants will not receive any training program from the research team. They only have their regular therapy from their own hospitals or clinics. The information of regular therapy, including the type, the frequency and the dosage, will be collected at T1, T2 and T3.

Intervention: The research team and independent therapists will ask caregivers to identify goals (before the first training session), and measure progress using goal-attainment scaling (GAS) at T1, T2 and T3 time points for the four groups. Two independent licensed occupational therapists (OTs) who will not involve the administration of assessments will provide the ROC-Stand training and conventional therapy programs, respectively. All participants in the 4 groups will continue their regular therapy from their own hospitals or clinics throughout the 24-week duration of the study, including physical therapy, occupational therapy, and speech therapy. All groups will receive the training program in the university for 2 hours/per session, 2 sessions/per week for a total of 12-week intervention. On licensed, independent OT will provide the ROC training programs and the other licensed, independent OT will provide the conventional therapy. The training programs for the two ROC training groups will be based on the ecological and dynamic systems theory. All the programs will be discussed by the family, the treating therapist and the research team. The programs for the two control group will be based on developmental and motor learning theories.

Follow-up: This period will involve a 12-week phase following the above treatment programs; during this time no treatment programs will be delivered to the participants except for their own regular therapy.

Data Reduction and Analysis: Social Looking and Interactions Measures: To examine participant's social looking and interactive behaviors, the following measures will be obtained via coding video footage during the 12-week intervention phase. Because young children, like adults, keep their eyes relatively centered in view most of the time. Thus, studies have been applied the center of the visual field to indicate the focus point. On the basis of these studies, the coding variables included face looking, body/toy/environment looking, child's and social partner's vocalizations, child-initiated and caregiver-initiated vocalizations/gesture, concurrent/overlapping vocalizations, conversation units and visual scan.

To compare the baseline characteristics of the major 2 groups categorized as mild and moderate motor delay, independent t-test (for data with normal distribution) and The Mann-Whitney U test (for data with non-normal distribution) will be conducted. Data will be analyzed based on an intention-to-treat analysis. A repeated measures analysis of variance (group [4] × time [3]) will be employed to evaluate the treatment effects on the primary and secondary outcomes among the 4 groups at T1, T2, and T3, followed by a post-hoc analysis using Bonferroni test to determine between which groups the differences occur.

For those data collected during the 12-week intervention, descriptive statistics (frequency, means, standard deviations) of social looking and interactions will be calculated and repeated measures analysis of variance (group [4] × time [12]) will be used to compare the effects among the 4 training groups during intervention. Furthermore, the quantitative data of energy expenditure and activity counts obtained from the ActiGraph® during intervention will be organized and calculated. A repeated measures analysis of variance (group [4] × time [12]) will also be used to compare the differences among the 4 groups. The mean frequency of total social looking and interactions will be calculated from the coding results of the 12-week intervention. SPSS 20.0 (SPSS Inc. Chicago, Illinois, USA) will be used for statistical analysis. Significance level will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. motor delays that resulted in motor impairments that prevented independent walking (standard deviation (SD) < -1.5, assessed by the Chinese Child Development Inventory (CCDI) via a pediatric physician)
2. can sit independently without support for 3 seconds
3. can stand independently for two seconds or to tolerate standing with support for 10 minutes
4. can reach for objects/toys with either one or two hands
5. the height is between 69 to 103 cm and the weight is between 7-18 kg
6. parents are able to provide consent for their child's participation in training programs

Exclusion Criteria:

1. children with severe sensory impairments such as blindness, deafness
2. the height is not between 69 to 103 cm and the weight is not between 7 to 18 kg
3. parents/caregivers are not able to make a time commitment for the training phase

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in General Mobility and Social Development at 12 weeks and 24 weeks as assessed by the Cinese version of Pediatric Evaluation of Disability Inventory (PEDI) | Assessment will occur 3 times during the whole study, including the first and last week of the 12-week intervention, and the end of the 12-week follow-up phase
  PEDI is a set of tests for children from 8 months to 6 years old. The PEDI quantified self-care, mobility, and social functions. The PEDI is especially useful for tracking changes in functional skills.
Social Looking and Interactions | The socialization behaviors will be followed for the duration of implementing the intervention phase, an expected average of 12 weeks.
  The behaviors of social looking and interactions are recorded from the head-mounted action cameras.The frequency and duration of the following will be coded: face looking, body looking, toy and environment looking, participants' and caregivers' vocalizations, child-initiated and caregiver-initiated vocalizations/gestures, concurrent/overlapping vocalizations, conversational units and visual scan.

SECONDARY OUTCOMES:
Physical Activity for Exploration as assessed by the number of counts recorded from the accelerators wearing on both wrists and the hip | The socialization behaviors will be followed for the duration of implementing the intervention phase, an expected average of 12 weeks.
  Each week the participant wears the accelerometers on both wrists and the hip during the 1 hour videotaping session, including 30-minute driving and 30-minute natural play. The accelerometers code the physical activity for driving and playing. Combining with the results from videotapes, this data enables us to understand the frequency and duration of bimanual use in different activities (i.e., manual exploration).
Change from baseline in General Development at 12 weeks and 24 weeks as assessed by The Bayley Scales of Development | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  An internationally recognized set of standardized developmental tests involves play and parental questionnaires. The Bayley has subsets of tests for motor (fine and gross), language (receptive and expressive), and cognitive development, ages from 0-3 years old.
Change from baseline in General Development at 12 weeks and 24 weeks as assessed by The Affordances in the Home Environment for Motor Development (AHEMD) | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  AHEMD is a reliable and valid assessment to assess the quality and quantity of motor development opportunities in the home during early childhood. Age-related AHEMD questionnaires were developed (3-to-18 months; and 18-to-42 months) and translated into four different languages: English, Chinese Portuguese, and Spanish. Test-retest reliabilities for AHEMD-Toddler-C were adequate (0.46~0.93). For convergent validity, the correlation coefficients between AHEMD and HOME were 0.44.
Change from baseline in Body Function/Structure at 12 weeks and 24 weeks as assessed by 5-repetition Sit-to-stand (STS) test | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  A test that measures the time require to complete five consecutive sit-to-stand to-sit cycle as quickly as possible timed using a stop watch. Participants will be tested barefoot on a firm mat and the starting position with hip flexed at 90 degree and knee flexed at 105 degree. The ICCs of intra-session reliability and test-retest reliability were 0.95 and 0.99 respectively. The convergent validity was supported by significant correlation with isometric muscle strength, scores of Gross Motor Function Measure, and gait function (r or rho = 0.45-0.78).
Change from baseline in Body Function/Structure at 12 weeks and 24 weeks as assessed by Revised Dimensions of Mastery Questionnaire (DMQ 18) - Chinese version | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  The Revised Dimensions of Mastery Questionnaire (DMQ 18) - Chinese version: was used to measure both instrumental and expressive aspects of mastery motivation by caregiver report. There are 7 scales (cognitive/object persistence, gross motor persistence, social mastery motivation with adults, social mastery motivation with children/peers, mastery pleasure, negative reactions to challenge in mastery situations, and general competence) and Likert-type items rated 1-5(from not at all like this child to exactly like this child). The DMQ 18 contained four parallel age-related versions for children aged 6 months to 19 years (infant, preschool, school-age rated by adults, and school-age self-report). The DMQ 18 show good internal consistency (.72-.96). The intra- and inter-rater reliability were acceptable for the DMQ18 (ICCs=0.61-0.87).
Change from baseline in Participation level at 12 weeks and 24 weeks as assessed by The Goal Attainment Scale (GAS) | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  GAS is a family-centered, criterion-referenced and responsive tool. There are 5 possible outcomes: a score of 0 means the child has attained the goal, whereas scores of -2 and -1 represent lower than expected performance and +1 and +2 are higher than expected performance. It has excellent inter-rater agreements with inter-class correlations of 0.90 or above. GAS was shown to correlate strongly with other measures that showed change, and it discriminated between lower and higher functional or QOL status.
Change from baseline in Parents' Perception at 12 weeks and 24 weeks as assessed by Parenting Stress Index (PSI) | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  PSI is a tool that was designed to measure the overall level of parenting stress experienced by parents of children between the ages of one month and twelve years. PSI showed very good reliability (from parent : .55-.80). The validity was well established (factorial validity: 41% of variance on child section accounted for by 6 factors; 44% on Parent section by 7 parent factors).
Change from baseline in Parents' Perception at 12 weeks and 24 weeks as assessed by self-developed questionnaires | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  A set of self-developed questionnaires from the previous studies will be revised and used at T1, T2 and T3 to examine parental perceptions on the training programs and children's capabilities

CONTACTS AND LOCATIONS:
Overall Officials: HsiangHan Huang, ScD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung University, Taoyuan, Taoyuan County, Taiwan